CLINICAL TRIAL: NCT06700551
Title: Evaluating the Efficacy of Mobile-Phone-Based Psychoeducation Intervention on Depression, Anxiety, and Stress in Dementia Caregivers
Brief Title: Mobile-Phone-Based Psychoeducation for Dementia Caregivers in Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nguyen Tran To Tran (Other)
Collaborators: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Sponsor-Investigator, Nguyen Tran To Tran, Lecturer, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 557-HDDD-DHYD
Record Dates: First submitted 2024-10-20; First posted 2024-11-22 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Depression, Anxiety; Stress
Keywords: dementia; caregiver; depression; anxiety; stress; intervention; psychoeducation; mobile-phone
MeSH Terms: conditions — Depression; Anxiety Disorders; Dementia

STUDY DESIGN:
Intervention Model Description: Psychoeducation
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducation Intervention Group (Experimental): In the intervention group, participants will receive interventions through the Zalo app on their mobile phones. Weekly, the investigator will send a topic for participants to learn about. Participants will have the opportunity to ask questions and share their feelings or experiences through the Zalo app.
  Interventions: Other: Psychoeducation
- Control group (No Intervention): Participants will receive usual care and will not receive any intervention

INTERVENTIONS:
Other: Psychoeducation — Each week, the investigator will send participants one topic through the chat function on the Zalo app. Before receiving the topic, participants will vote on which topic they would like to learn about. The topics will be presented as videos and will cover the following seven areas: providing everyday care, being a caregiver, self-care, knowledge about dementia, fall prevention, pressure injury prevention and care, and managing behavior changes.They may ask questions related to providing dementia care or share their feelings via the chat on the Zalo app.
  Arms: Psychoeducation Intervention Group

SUMMARY:
The goal of this study is to determine whether a mobile phone-based psychoeducational intervention can reduce stress among caregivers of individuals with dementia in Vietnam. The primary research question is: Does the intervention reduce levels of depression, anxiety, and stress among participants? The secondary research question is: Does the intervention increase caregivers' knowledge about dementia, enhance social support, or reduce caregiver burden?

DETAILED DESCRIPTION:
The study consists of two groups: an intervention group and a control group. Participants in the intervention group will receive psychoeducational content through the Zalo app on their mobile phones. Weekly, they will be provided with a topic related to dementia care, such as daily caregiving, fall prevention, pressure injury prevention and care, self-care, and coping as a caregiver. Levels of depression, anxiety, and stress will be assessed both before and after the intervention. In the control group, participants will continue receiving standard care.

ELIGIBILITY:
Inclusion Criteria:

* Primary Caregiver Requirement: Participants must have been the primary caregivers of poeple with dementia for at least the past 6 months and plan to continue in this role for the next 6 months of the intervention. Patients with demeentia criteria: Patients must have been diagnosed with dementia for at least 6 months and reside within the community.
* Language and Education Requirement: Participants must be able to read and understand Vietnamese (with at least a primary education level) and be willing to participate in the study.
* Smartphone Requirement: Participants must own a smartphone with the Zalo app or be willing to install it (with a brief training session provided for new users).
* Age Requirement: Participants must be aged 18 years or older.

Exclusion Criteria:

* Having any acute diseases or cognitive impairment (screening by Mini-Cog) or
* Having vision or hearing impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2024-10-26 (Actual); Primary Completion 2025-07-05 (Actual); Study Completion 2025-07-05 (Actual)

PRIMARY OUTCOMES:
Depression, anxiety and stress levels | The evaluation period will span from enrollment to the end of the 7-week intervention and continue through three months post-intervention. Assessments will be conducted at three key time points: baseline (prior to the intervention), immediately after the
  Levels of depression, anxiety, and stress will be assessed using the Depression, Anxiety, and Stress Scale (DASS-21), which includes three subscales. Each subscale has a scoring range from 0 to 42, resulting in a total possible score between 0 and 126. Higher scores indicate more severe symptoms and worse outcomes.

SECONDARY OUTCOMES:
Demetia knowledge | The evaluation period will extend over 9 months. Assessments will be conducted at three time points: baseline (before the intervention), immediately post-intervention, and three months post-intervention.
  Participants' demntia knowledge will be assessed using a questionnaire adapted from the Northern Ireland Life and Times Survey, consisting of 7 items. The total score ranges from 0 to 7, with higher scores indicating better knowledge and understanding of dementia.
Caregiver burden | The evaluation period will extend over 9 months. Assessments will be conducted at three key time points: baseline (before the intervention), immediately post-intervention, and three months post- intervention.
  Participants will be assessed using the Zarit 4-Item Burden Interview, which consists of four items. Each item is rated on a scale of 1 to 4, with higher scores indicating a greater sense of caregiver burden.
Percieved social support | The evaluation will span 9 months, with assessments conducted at three key points: baseline (before the intervention), immediately post-intervention, and three months post-intervention.
  Participants will be assessed using the Multidimensional Perceived Social Support Scale (MSPSS), which consists of 12 items. Each item is rated on a 7-point Likert scale, ranging from 1 (very strongly disagree) to 7 (very strongly agree). The total score ranges from 12 to 84, with higher scores indicating greater levels of perceived social support.

CONTACTS AND LOCATIONS:
Overall Officials: Tran TT Nguyen, MD, MSc, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- Nhan Dan Gia Dinh Hospital, Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No
To ensure participant confidentiality, study results will only be shared upon the request and with the explicit agreement of the principal investigator.

REFERENCES:
- [Result] Bruwer B, Emsley R, Kidd M, Lochner C, Seedat S. Psychometric properties of the Multidimensional Scale of Perceived Social Support in youth. Compr Psychiatry. 2008 Mar-Apr;49(2):195-201. doi: 10.1016/j.comppsych.2007.09.002. Epub 2007 Dec 21. PMID 18243894
- [Result] McParland P, Devine P, Innes A, Gayle V. Dementia knowledge and attitudes of the general public in Northern Ireland: an analysis of national survey data. Int Psychogeriatr. 2012 Oct;24(10):1600-13. doi: 10.1017/S1041610212000658. Epub 2012 May 17. PMID 22591515
- [Derived] Nguyen TTT, Vu LDT, Nguyen TC, Truong KT, Thai TT, Than THN, Nguyen HT. Mobile App Psychoeducation for Dementia Caregivers In Vietnam: A Randomized Controlled Trial. J Multidiscip Healthc. 2025 Oct 23;18:6871-6885. doi: 10.2147/JMDH.S557573. eCollection 2025. PMID 41158517
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/22591515/
- See also: https://pubmed.ncbi.nlm.nih.gov/18243894/ — https://pubmed.ncbi.nlm.nih.gov/18243894/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/7726811/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/11574710/